CLINICAL TRIAL: NCT01237132
Title: EAST-WEST HEPATOCELLULAR CARCINOMA STUDY GROUP
Status: Completed | Type: Observational
Sponsor: University of Milan (Other)
Responsible Party: GUIDO TORZILLI MD, PHD, UNIVERSITY OF MILAN
Other Study IDs: HCC EWE
Record Dates: First submitted 2010-11-08; First posted 2010-11-09 (Estimated); Last update posted 2010-11-09 (Estimated); Status verified 2009-12

CONDITIONS: Carcinoma, Hepatocellular
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The current treatment guidelines of hepatocellular carcinoma (HCC) of the American and European Associations for the Study of Liver Disease are based on the Barcelona-Clinic-Liver-Cancer classification (BCLC), which does not recommend surgery in patients with large, multinodular and macrovascular invasive disease. The aim of this study was to investigate the role of hepatic resection in a large retrospective multicentric cohort of patients resected for HCC regardless of the BCLC indications.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of hepatocellular carcinoma
* candidate to liver resection as a curative treatment

Exclusion Criteria:

* uncertain diagnosis of hepatocellular carcinoma
* uncertain follow-up data

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients affected by HCC
Sampling Method: Non-Probability Sample

PRIMARY OUTCOMES:
Overall survival of resected patients for HCC
  The primary endpoint of the study was the overall survival of patients resected for HCC in any stage of the BCLC classification.

SECONDARY OUTCOMES:
Disease-free survival of resected patients for HCC
  The secondary endpoint was the disease-free survival of patients resected for HCC among the BCLC stages.